CLINICAL TRIAL: NCT06728527
Title: PartBreCon-Pro Study: PARTial BREast RECONstruction With Chest Wall Perforator Flap, a PROspective Study of Clinical and Patient Reported Outcomes
Brief Title: PARTial BREast RECONstruction With Chest Wall Perforator Flap
Acronym: PartBreCon
Status: Recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Amit Agrawal, Consultant Oncoplastic Breast Surgeon, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: ID5342
Record Dates: First submitted 2024-11-26; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Breast Carcinoma; Breast Neoplasms; Breast Surgery; Breast Reconstruction Surgery
Keywords: breast oncoplastic, recon, chest wall perforator flap, PROMS
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to ascertain the outcomes following partial breast reconstruction using chest wall perforator flaps after breast conservation surgery.

DETAILED DESCRIPTION:
The Main Outcomes and Measures are:

A) Patient Demographics and Tumour characteristics

1. Patient demographics: age, body mass index (BMI), comorbidities
2. Preoperative tumour characteristics and location influencing surgical planning

B) Treatment characteristics

1. Surgical: operative data, including flap types and distribution
2. Oncological: systemic therapies (adjuvant and neoadjuvant), radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing partial breast reconstruction using CWPF for primary breast cancer
* Delayed correction of breast deformity following previous BCS
* Each surgeon is to have performed a minimum of 10 CWPFs
* Each centre anticipates completing a minimum of 10/year

Exclusion Criteria:

* Patients undergoing volume displacement BCS
* Patients undergoing mastectomy +/- immediate breast reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancers
Study Population: Women over the age of 18 years who would have been offered all options (simple wide local excision, therapeutic mammaplasty, mastectomy with or without immediate whole breast reconstruction)
Sampling Method: Probability Sample
Enrollment: 1001 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Surgical Complications | Within 30 days of surgery
  Outcomes:
  • Rates of complications (e.g., Haematoma, Seroma, Infection, Delayed Wound healing, Fat necrosis, Flap loss, etc).
  Measures:
  • Complication rates stratified by severity (e.g., Clavien-Dindo classification).

SECONDARY OUTCOMES:
Oncological Clearance | From enrolment until the date of re-operation within 12 months of first surgery, or the end of study, whichever came first.
  Outcomes:
  • Effectiveness of surgery in achieving oncological goals.
  Measures:
  • Re-operation rates: Proportion of patients requiring further surgery (re-excisions and/or mastectomy) to achieve Oncological clearance.
Revisional surgery | From enrolment until the date of revision within 36 months of surgery, or the end of study, whichever came first.
  Outcomes:
  • Frequency and reasons for additional surgical procedures.
  Measures:
  • Revision rates by indication (e.g., aesthetic concerns, complication management).
Oncological: Recurrence | From enrolment until the date of recurrence, or the end of study, whichever came first, assessed up to 36 months
  Outcomes:
  • Recurrence rates (local, regional, distant).
  Measures:
  • Time to recurrence (mean/median in months).
Oncological: Survival | From enrolment until the date of death, or the end of study, whichever came first, assessed up to 36 months
  Outcomes:
  • Survival rates
  Measures:
  • Disease-free survival (DFS) and overall survival (OS) (mean/median in months).

OTHER OUTCOMES:
Patient-reported outcomes: Patient satisfaction and quality of life | Pre-operative, Post-operative and Post-radiotherapy (6 months).
  Outcomes:
  • Patient satisfaction and quality of life (QoL).
  Measures:
  • Measurement using a validated instrument, BREAST-Q, which converts the individual patient response items into a BREAST-Q score ranging from 0-100; a higher score means greater satisfaction of better QoL
Patient-reported outcomes: Upper extremity dysfunction | Pre-operative, Post-operative and Post-radiotherapy (6 months).
  Outcomes:
  • Disability of the Arm, Shoulder and Hand
  Measures:
  • Measurement using a validated instrument, QuickDASH (an abbreviated version of the Disability of the Arm, Shoulder, and Hand), which converts the individual patient response items into a QuickDASH score ranging from 0 to 100; a higher score means a greater level of disability and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Agrawal, Principal Investigator — Cambridge University Hospitals NHS Trust
Locations (1):
- Cambridge University Hospitals NHS Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Since it is a large international observational study, any sharing will need approval from all though anonymised data might be shareable (to be decided later).

REFERENCES:
- [Background] Agrawal A, Romics L, Thekkinkattil D, Soliman M, Kaushik M, Barmpounakis P, Mortimer C, Courtney CA, Goyal A, Garreffa E, Carmichael A, Lane RA, Rutherford C, Kim B, Achuthan R, Pitsinis V, Goh S, Ray B, Grover K, Vidya R, Murphy J; PartBreCon Collaborators. 'PartBreCon' study. A UK multicentre retrospective cohort study to assess outcomes following PARTial BREast reCONstruction with chest wall perforator flaps. Breast. 2023 Oct;71:82-88. doi: 10.1016/j.breast.2023.07.007. Epub 2023 Jul 17. PMID 37544090
- [Background] Garreffa E, Meattini I, Coles CE, Agrawal A. Use of tumour bed boost radiotherapy in volume replacement oncoplastic breast surgery: A systematic review. Crit Rev Oncol Hematol. 2023 Jun;186:103996. doi: 10.1016/j.critrevonc.2023.103996. Epub 2023 Apr 14. PMID 37061072
- [Background] Agrawal A. Oncoplastic breast surgery and radiotherapy-Adverse aesthetic outcomes, proposed classification of aesthetic components, and causality attribution. Breast J. 2019 Mar;25(2):207-218. doi: 10.1111/tbj.13193. Epub 2019 Feb 1. PMID 30710399
- [Background] Association of Breast Surgery A. NHSBSP and ABS Audit. Accessed 24.05.2020, https://associationofbreastsurgery.org.uk/professionals/audit/nhs-breast-screening-programme-audit/
- [Background] Garreffa E, Hughes-Davies L, Russell S, Lightowlers S, Agrawal A. Definition of Tumor Bed Boost in Oncoplastic Breast Surgery: An Understanding and Approach. Clin Breast Cancer. 2020 Aug;20(4):e510-e515. doi: 10.1016/j.clbc.2020.03.003. Epub 2020 Mar 20. PMID 32284305
- [Background] Agrawal A, Mirshekar-Syahkal B. Use of combination of modules of BREAST-Q in partial breast reconstruction with lateral chest wall perforator flap. Eur J Surg Oncol. 2016;42(5):S39. doi:https://doi.org/10.1016/j.ejso.2016.02.155
- [Background] Navin C, Agrawal A, Kolar KM. The use of latissimus dorsi miniflap for reconstruction following breast-conserving surgery: experience of a small breast unit in a district hospital. World J Surg. 2007 Jan;31(1):46-50. doi: 10.1007/s00268-006-0396-7. PMID 17180559
- [Background] Hamdi M, Van Landuyt K, Monstrey S, Blondeel P. Pedicled perforator flaps in breast reconstruction: a new concept. Br J Plast Surg. 2004 Sep;57(6):531-9. doi: 10.1016/j.bjps.2004.04.015. PMID 15308400
- [Background] Roy PG, Tenovici AA. Staged approach to partial breast reconstruction to avoid mastectomy in women with breast cancer. Gland Surg. 2017 Aug;6(4):336-342. doi: 10.21037/gs.2017.03.08. PMID 28861373
- [Background] Brouwers PJAM, van Werkhoven E, Bartelink H, Fourquet A, Lemanski C, van Loon J, Maduro JH, Russell NS, Scheijmans LJEE, Schinagl DAX, Westenberg AH, Poortmans P, Boersma LJ; Young Boost Trial research group. Predictors for poor cosmetic outcome in patients with early stage breast cancer treated with breast conserving therapy: Results of the Young boost trial. Radiother Oncol. 2018 Sep;128(3):434-441. doi: 10.1016/j.radonc.2018.06.020. Epub 2018 Jul 3. PMID 29980320
- See also: Lead Site — https://www.cuh.nhs.uk/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT06728527/Prot_SAP_000.pdf